CLINICAL TRIAL: NCT02342015
Title: Effect of Atorvastatin on OPG/RANK/RANKL Expression in Immune Cells and Circulating Levels of Osteoprogenitor Cells
Brief Title: Effect of Atorvastatin on Bone-vascular Axis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Marcello Rattazzi, Assistant Professor, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Studio clinico n° 14/AULSS 9
Record Dates: First submitted 2014-11-28; First posted 2015-01-19 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Osteoporosis; Hypercholesterolemia
MeSH Terms: conditions — Osteoporosis; Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atorvastatin (Experimental): Atorvastatin 40 mg/day for three months
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 40mg/day for three months
  Other Names: Lipitor

SUMMARY:
Background: Circulating osteoprogenitors and RANKL expression in immune cells have been implicated in the pathogenesis of osteoporosis and vascular calcification. The role played by statin therapy in the bone-vascular axis is unknown.

Methods: Twenty naïve post-menopausal osteoporotic hypercholesterolemic women will be treated with Atorvastatin 40 mg/day for three months. Blood samples will be collected at baseline and at the end of the treatment. Gene expression analysis will be performed to assess modification in OPG/RANK/RANKL expression in isolated T-cells and monocytes. A flow cytometry analysis will be used to study changes in the levels of circulating osteoprogenitor cells.

DETAILED DESCRIPTION:
Background: A considerable number of clinical studies have shown that osteoporosis carries a signiﬁcant increase in cardiovascular risk. Although the pathophysiological substrate of the so-called bone-vascular axis is still elusive, an important role is attributed to the OPG/RANK/RANKL triad, a master regulator of bone remodeling. In addition, circulating osteoprogenitors have been recently described as a new subset of immature cells harbouring pro-calciﬁc potential in the vasculature and heart valves. Nevertheless, a number of studies indicated that the accumulation of lipid oxidation products within the skeleton may contribute to pathological bone resorption, mainly through the inhibition of osteoblast differentiation and the induction of osteoclast maturation/activation. Starting from these notions, we sought to investigate whether treatment with Atorvastatin can affect circulating levels of osteo-progenitor cells and OPG/RANK/RANKL expression in T cells and monocytes in hypercholesterolemic postmenopausal osteoporotic women.

Methods: We will enrol 20 consecutive hypercholesterolemic (LDL-C ≥130 mg/dL) women with newly diagnosed osteoporosis who refer to the Osteoporosis and Bone Metabolism Unit of the Cà Foncello Hospital in Treviso. Diagnosis of osteoporosis was based on T-score ≤2.5 SD at either the lumbar spine or femoral neck. All patients will receive Atorvastatin 40 mg/day for 3 months. Blood samplings will be performed at the time of enrolment and at the end of the treatment period. During the study, the patients will not be treated with calcium, vitamin D, and bisphosphonates. We will exclude women with clinical judgment of high risk of bone fracture. At the beginning of the study and after 3 months, serum samples will be collected to assess the lipid proﬁle (total cholesterol [TC], LDL-C, HDL-C, triglycerides [TG]), level of hs-CRP, osteocalcin (OCN), bone alkaline phosphatase (BAP), cross-linked carboxy-terminal telopeptide of type I collagen (CTX-I), and OPG. Blood samples at enrolment and after three months will be also obtained to quantify circulating osteoprogenitor cells (flow cytometry) and gene expression of OPG/RANK/RANKL in mononuclear cells (RT-PCR).

Flow cytometry analysis (FACS): identiﬁcation and quantiﬁcation of circulating osteoprogenitor cells will be performed using polychromatic ﬂow cytometry. Brieﬂy, after red blood cell lysis, peripheral blood progenitor cells will be analysed for the surface expression of CD34, OCN and BAP using Fitc-conjugated anti-human CD34, PE-conjugated anti-human OCN, and APC-conjugated anti-human BAP.

Gene expression analysis: pure and viable monocytes and T cells will be obtained from blood samples by negative isolation using Dynabeads Untouched Human Monocytes and Dynabeads Untouched Human T cells respectively. Total RNA from both cell types will be collected using and stored at -80°Cuntil analysis. The levels of RANK, RANKL, and OPG transcripts will be then quantiﬁed by real-time PCR .

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed osteoporosis (T score ≤ -2.5 SD at either the lumbar spine or femoral neck)
* LDL-cholesterol ≥ 130 mg/dl

Exclusion Criteria:

* History of bone fractures,
* Clinical evidence of atherosclerotic disease
* CKD (stage III-V),
* Liver disease
* COPD
* Rheumatic disorders;
* Current or previous treatment with statins, steroids, hormonal replacement therapies, and antiosteoporotic drugs (including vitamin D and calcium supplementation)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Rattazzi, MD, Principal Investigator — University of Padova, Department of Medicine

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atorvastatin
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Atorvastatin
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 20
Total Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 257.7 (24.1)
high-sensitivity C-reactive protein (hs-CRP) [Median (Inter-Quartile Range); unit: mg/dl] | 1 [0.64 to 1.81]
Osteocalcin (OCN) [Mean (Standard Deviation); unit: ng/ml] | 25.4 (5.7)
Bone Alkaline Phosphatase (BAP) [Mean (Standard Deviation); unit: mcg/L] | 14.5 (2.5)
Osteoprotegerin (OPG) [Mean (Standard Deviation); unit: pg/ml] | 644.5 (271.8)
cross-linked carboxy-terminal telopeptide of type I collagen-I (CTX-I) [Mean (Standard Deviation); unit: ng/ml] | 529.3 (178.6)
Calcium [Mean (Standard Deviation); unit: mmol/L] | 2.36 (0.06)
Phosphorus [Mean (Standard Deviation); unit: mmol/L] | 1.13 (0.10)
Vitamin D3 [Mean (Standard Deviation); unit: nmol/L] | 74.8 (45.9)
CD34+/BAP+ cells [Mean (Standard Deviation); unit: cells/million events] | 136.1 (28.9)
CD34+/OCN+ cells [Mean (Standard Deviation); unit: cells/million events] | 200.9 (40.8)
OCN+/BAP+ cells [Mean (Standard Deviation); unit: cells/million events] | 11180.2 (3657.3)
CD34+/OCN+/BAP+ cells [Mean (Standard Deviation); unit: cells/million events] | 123.6 (29.5)

OUTCOME MEASURES:

1. Primary Outcome: Relative Change in OPG/RANK/RANKL mRNA Expression in Isolated T Cells and Monocytes
Description: Isolated T cells and monocytes will be obtained at baseline and at the end of the treatment period. Gene expression analysis will be performed in each cell type to assess the expression level of OPG, RANK, and RANKL at baseline and after three months of treatment.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: relative fold change
Arm/Group | Atorvastatin
Number analyzed (Participants) | 20
relative fold change | 0.76 (0.1)
Statistical Analysis 1: Comparison: Atorvastatin; Test type: Other; p < 0.05, wilcoxon signed-rank test

2. Primary Outcome: Change in Circulating Levels of Osteoprogenitor Cells (CD34+/OCN+/BAP+ Cells)
Description: Circulating levels of osteoprogenitor cells (CD34+/OCN+/BAP+ cells) will be measured by FACS analysis in each patient at baseline and after three months of treatment with Atorvastatin.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: cells/million events
Arm/Group | Atorvastatin
Number analyzed (Participants) | 20
cells/million events | 59.1 (13.6)
Statistical Analysis 1: Comparison: Atorvastatin; Test type: Other; p < 0.05, paired Student's t-test

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No